CLINICAL TRIAL: NCT02246946
Title: Efficacy of the Addition of Positive Airway Pressure to Conventional Chest Physiotherapy in the Time to Resolution of Pleural Effusion After Drainage
Brief Title: Positive Airway Pressure on Pleural Effusion After Drainage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Adriana Claudia Lunardi, Professor on Master's and Doctoral Programs in Physical Therapy of Universidade Cidade de São Paulo, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNICID14
Record Dates: First submitted 2014-09-16; First posted 2014-09-23 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; chest tube; respiratory therapy; intermittent positive-pressure breathing; lung function; pulmonary complications
MeSH Terms: conditions — Pleural Effusion | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Positive Airway Pressure group (Experimental): The patients allocated to this group will undergo bronchial hygiene treatments administered with a high-frequency oscillator for 5 sets of 10 repetitions, lung expansion exercises using flow oriented incentive spirometry for 5 sets of 20 repetitions and walking for 100 meters (i.e., the same treatment that will be administered to the Conventional Chest Physiotherapy group). Additionally, this group will receive positive airway pressure breathing with 15 mmHg by a device via a rubber facial mask for 30 minutes in a sitting position.
  Interventions: Device: Positive Airway Pressure
- Conventional Chest Physiotherapy group (Active Comparator): In the sitting position, the patients allocated to this group will undergo bronchial hygiene treatments administered with a high-frequency oscillator for 5 sets of 10 repetitions, lung expansion exercises using flow oriented incentive spirometry for 5 sets of 20 repetitions and positive airway pressure breathing with 4 mmHg via a rubber facial mask for 5 minutes in a sitting position. These patients will also walk for 100 meters.
  The use of positive pressure breathing with 4 mmHg has no therapeutic value, but will help keep the blinding of assessors by the presence of the equipment in the room and mark the patient's skin.
  Interventions: Other: Conventional Chest Physiotherapy
- Control group (Placebo Comparator): The patients allocated to this group will receive positive airway pressure breathing with 4 mmHg (without therapeutic value) via a rubber facial mask for 30 minutes in a sitting position.
  The use of positive pressure breathing with 4 mmHg has no therapeutic value, but will help keep the blinding of assessors by the presence of the complete kit of equipment in the room.
  Interventions: Procedure: Control group

INTERVENTIONS:
Device: Positive Airway Pressure — To this group, Intermittent Positive Airway Pressure Breathing with 15 mmHg by Muller Reanimatior (Engemed, Brazil) device with a rubber facial mask will be provide
  Arms: Positive Airway Pressure group
Other: Conventional Chest Physiotherapy — To this group, routine physiotherapy exercises will be conducted plus Intermittent Positive Airway Pressure Breathing with 4 mmHg by Muller Reanimatior (Engemed, Brazil) device with a rubber facial mask will be provide
  Arms: Conventional Chest Physiotherapy group
Procedure: Control group — to this group, Airway Pressure Breathing with 4 mmHg by Muller Reanimatior (Engemed, Brazil) device with a rubber facial mask will be provide
  Arms: Control group

SUMMARY:
The purpose of this study is to determine if the addition of intermittent positive airway pressure breathing (specific lung expansion technique) to conventional chest physiotherapy chest drainage is effective to accelerate the reabsorption of pleural effusion and consequently decrease the duration of chest tube drainage and respiratory system impairment. These effects would decrease hospital stay lengths and the incidence of pulmonary complications.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* presence of pleural effusion
* have undergone chest drain for fewer than 24 hours

Exclusion Criteria:

* contraindication to the use of non-invasive equipment that generates positive airway pressure (such as: intolerance, phobia, drowsiness, restlessness, confusion, hemodynamic instability requiring vasopressor therapy, systolic blood pressure < 90 mmHg, facial trauma, ineffective cough or inability to swallow, nausea or vomiting, upper gastrointestinal bleeding, acute myocardial infarction within the last 48 hours, pneumothorax or bullous emphysema)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2014-12; Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Duration of chest tube drainage | All patients will be followed for the duration of hospital stay, an expected average of 7 days of chest drainage
  The criteria for the removal the chest drain will an output of transudative fluid over 24h ≤ 200 ml and full lung expansion on chest radiography

SECONDARY OUTCOMES:
Spirometry | On the 4th and 8th days after the beginning of the intervention protocol. Or on the day of hospital discharge if it occurs prior to the 8th day of protocol
  The blind assessor will use a portable spirometer according previously established implementation and acceptability criteria. The following variables will be considered: forced vital capacity, forced expiratory volume in the 1st second, and forced expiratory flow between 25% and 75% of the curve. The predictive values for the Brazilian population will be used
Peripheral Oxygen Saturation | On the 4th and 8th days after the beginning of the intervention protocol. Or on the day of hospital discharge if it occurs prior to the 8th day of protocol
  The patients will be required to breath room air (without supplemental oxygen) for at least 10 minutes prior to the assessments. The blind assessor will use a portable pulse oximeter.
Pulmonary complications | All patients will be followed for the duration of hospital stay, an expected average of 10 days
  The occurrence of the following complications will be monitored until the day of hospital discharge by a physician blinded to the intervention groups: pneumonia (chest radiography with pulmonary infiltrate associated with two of the following signs: purulent expectoration, temperature above 38.3°C and a greater than 25% increase in baseline leukocyte count with hyperthermia); atelectasis (RX associated with abnormal chest acute respiratory symptoms); and hypoxemia (peripheral oxygen saturation associated with respiratory symptoms below 85%)
Length of hospital stay | All patients will be followed for the duration of hospital stay, an expected average of 10 days
  The number of days in the hospital after chest drainage until discharge will be counted for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Adriana C Lunardi, PhD, Study Director — Universidade Cidade de Sao Paulo; Elinaldo C Santos, MSc, Principal Investigator — Hospital das Clínicas Dr. Alberto Lima
Locations (1):
- Hospital das Clínicas Dr. Alberto Lima, Macapá, Amapá, Brazil

REFERENCES:
- [Derived] Dos Santos EDC, da Silva JS, de Assis Filho MTT, Vidal MB, Monte MC, Lunardi AC. Adding positive airway pressure to mobilisation and respiratory techniques hastens pleural drainage: a randomised trial. J Physiother. 2020 Jan;66(1):19-26. doi: 10.1016/j.jphys.2019.11.006. Epub 2019 Dec 13. PMID 31843426
- [Derived] da Conceicao Dos Santos E, Lunardi AC. Efficacy of the addition of positive airway pressure to conventional chest physiotherapy in resolution of pleural effusion after drainage: protocol for a randomised controlled trial. J Physiother. 2015 Apr;61(2):93. doi: 10.1016/j.jphys.2014.11.016. Epub 2015 Mar 3. PMID 25744852